CLINICAL TRIAL: NCT04528329
Title: Anosmia and / or Ageusia in COVID-19: Timeline, Treatment With Early Corticosteroid and Recovery
Brief Title: Anosmia and / or Ageusia and Early Corticosteroid Use
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ClinAmygate (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR0013
Record Dates: First submitted 2020-08-24; First posted 2020-08-27 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Covid19; Anosmia
MeSH Terms: conditions — COVID-19; Anosmia | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early CS (Experimental): early use of dexamethasone as early as the laboratory confirmation of inflammation.
  Interventions: Drug: Early-Dexamethasone
- Late CS (Active Comparator): Dexamethasone is to be used lately upon the deterioration of cases
  Interventions: Drug: Late dexamethazone

INTERVENTIONS:
Drug: Early-Dexamethasone — early use of dexamethasone as early as laboratory evidence of high inflammatory markers
  Other Names: Dexamethasone
  Arms: Early CS
Drug: Late dexamethazone — Use of dexamethasone on deterioration of the cases with increased severity
  Other Names: Dexamethasone
  Arms: Late CS

SUMMARY:
Time to recover of Anosmia and / or ageusia and early corticosteroid use

DETAILED DESCRIPTION:
In a study of dexamethasone kinetics in two groups of 15 patients with community-acquired pneumonia, one group was treated with dexamethasone 6 mg/day by mouth and the other with 4 mg/day intravenously. The apparent volume of distribution was 1 L/kg in both groups, but the half-life after oral administration was approximately 7 hours, and after intravenous administration 9 hours. The bioavailability of oral dexamethasone was 81% (95% CI = 54-121%). However, the biological half-life of dexamethasone is much longer, of the order of 36-54 h compared with 18-36 h for prednisolone.

Time to recover of Anosmia and / or ageusia and early corticosteroid use

ELIGIBILITY:
Inclusion Criteria:

* Any case with COVID-19
* Age more than or equal to 18 years
* Mild to moderate severity

Exclusion Criteria:

* Diabetes
* Any contra-indication for the interventional drug
* Mentally disabled cases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-03-30 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Time to recovery | one to 6 weeks
  Time to recovery from anosmia and / or agusia

CONTACTS AND LOCATIONS:
Overall Officials: Emad R Issak, MD, Study Director — Assalam Clinics
Locations (1):
- Asalam, Maadi, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spoorenberg SM, Deneer VH, Grutters JC, Pulles AE, Voorn GP, Rijkers GT, Bos WJ, van de Garde EM. Pharmacokinetics of oral vs. intravenous dexamethasone in patients hospitalized with community-acquired pneumonia. Br J Clin Pharmacol. 2014 Jul;78(1):78-83. doi: 10.1111/bcp.12295. PMID 24400953